CLINICAL TRIAL: NCT04407715
Title: The Effect Of Minimal and High Flow Anesthesia on Optic Nerve Sheath Diameter in Laparotomic Gynecological Surgery
Brief Title: Anesthesia on Optic Nerve Sheath Diameter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Anıl Onur, Principle İnvestigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018/11-0
Record Dates: First submitted 2020-03-10; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Optic Nerve Sheath Diameter
Keywords: Minimal Flow Anesthesia; Optic Nerve Sheath Diameter

STUDY DESIGN:
Intervention Model Description: A total of 80 patients who underwent laparotomic gynecological surgery were divided into two groups prospectively: high flow of 2 L/min and minimal flow of 0.5 L/min. Anesthesia was maintained with 50% oxygen-50% air at 2 L/min and desflurane at 1.1 MAC in Group 1 (n=40) and with 50% oxygen-50% air at 2 L/min and desflurane at 1.1 MAC in Group 2 (n=40). After 10-15 minutes, group 2 was administered minimal flow with 50-60% oxygen-40-50% air at 0.5 L/min and desflurane, and 10 minutes before the end of the surgery, the patients were switched to high flow with 50% oxygen-50% air at 2 L/min.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Flow Anesthesia, Low Flow Anesthesia (Placebo Comparator): . The patients were randomly allocated to one of the two groups of fresh gas flows using the closed-envelope technique: 2 L/min high flow and 0.5 L/min minimal flow. Group 1 (n = 40) was operated under high flow anesthesia with 50% O2 - 50% air at 2 L/min and desflurane at 1.1 MAC for the duration of the surgery. For anesthesia maintenance, Group 2 (n=40) was administered 50% oxygen - 50% air at 2 L/min and desflurane for 10-15 minutes. After reaching 1.1 MAC, it was switched to minimal flow with 50-60% oxygen- 40-50% air at 0.5 L/min and desflurane. 10 minutes before the end of the surgery, it was switched to high flow with 50% oxygen -50% air at 2 L/min.
  Interventions: Procedure: The Effect Of Minimal and High Flow Anesthesia on Optic Nerve Sheath Diamater
- Peroperetive Optic Nerve Sheath Diameter (Active Comparator): Optic nerve sheath diameter measurements were performed by an experienced and the same anesthetist. In the measurements, the GE Healthcare Logiq e series USG device and 12-MHz linear probe were used. Longitudinal and transverse axis images were obtained on both eyelids while the patient was in the supine position. Measurements were taken 3 mm behind the optic nerve head
  Interventions: Procedure: The Effect Of Minimal and High Flow Anesthesia on Optic Nerve Sheath Diamater

INTERVENTIONS:
Procedure: The Effect Of Minimal and High Flow Anesthesia on Optic Nerve Sheath Diamater — The patients were randomly allocated to one of the two groups of fresh gas flows using the closed-envelope technique: 2 L/min high flow and 0.5 L/min minimal flow.

SUMMARY:
Different amounts of anesthetic gas can be used in the obstetric gynecological surgery operations to be performed with open method. Researchers aimed to compare the effect of gas changes on intraocular nerve diameter by ultrasonography.

DETAILED DESCRIPTION:
A total of 80 patients who underwent laparotomic gynecological surgery were divided into two groups prospectively: high flow of 2 L/min and minimal flow of 0.5 L/min. Anesthesia was maintained with 50% oxygen-50% air at 2 L/min and desflurane at 1.1 MAC in Group 1 (n=40) and with 50% oxygen-50% air at 2 L/min and desflurane at 1.1 MAC in Group 2 (n=40). After 10-15 minutes, group 2 was administered minimal flow with 50-60% oxygen-40-50% air at 0.5 L/min and desflurane, and 10 minutes before the end of the surgery, the patients were switched to high flow with 50% oxygen-50% air at 2 L/min.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* ASA I-II
* Who underwent laparotomic gynecological surgery

Exclusion Criteria:

* Patients with obstructive pulmonary disease
* Patients with decompensated diabetes, those with a fasting period of more than 12 hours -Acute alcohol intoxication
* Chronic alcohol use
* Who refuse to participate in the study
* Who are not cooperative, do not speak Turkish
* Who had known eye disease (glaucoma, retinal detachment), had a previous history of eye surgery,
* Increased intracranial pressure findings (intracranial lesion, previous cerebrovascular diseases
* Body mass index of > 40kg/m2
* ASA > III

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Optic Nerve Sheath Diamater | 2 hours operation time
  Optic nerve sheath diamater measurements of the patients were recorded before and during the surgery at specified time points (T0: awake, T1: High fresh gas flow after induction at the 10th min., T2: Inhalation anesthesia at the 30th min., T3: Inhalation anesthesia at the 60th min., T4: Inhalation anesthesia at the 90th min., T5: Before extubation).A typical optic nerve sheath is generally less than 5 mm in diameter, and diameters greater than 5.5 mm predict an ICP of ≥20 cm H2O with 100% sensitivity and specifity

SECONDARY OUTCOMES:
Peroperative Complications | 2 hours operation time
  Complications during the surgery (decreased oxygen levels, hypercapnia, hypotension, hypertension, bradycardia, tachycardia, rhythm disorders) were recorded.
Postoperative Complications | postop 20 minutes
  Complications in the recovery room (respiratory distress, decreased oxygen levels, hypotension, hypertension, bradycardia, tachycardia, vomiting, rhythm disorders) were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Anıl Onur, MD, Principal Investigator — University of Health Science Bursa Yüksek Ihtisas Training and Research Hospital; H.Erkan Sayan, MD, Study Director — University of Health Science Bursa Yüksek Ihtisas Training and Research Hospital; Tugba Onur, MD, Study Chair — University of Health Science Bursa Yüksek Ihtisas Training and Research Hospital; Umran Karaca, MD, Study Chair — University of Health Science Bursa Yüksek Ihtisas Training and Research Hospital; Canan Yılmaz, MD, Study Chair — University of Health Science Bursa Yüksek Ihtisas Training and Research Hospital
Locations (1):
- University of Health Sciences Bursa Yüksek İhtisas Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No